CLINICAL TRIAL: NCT00574899
Title: Multi-Institutional Inter-SPORE Prostate Biomarker Study
Brief Title: Prostate Biomarker Study
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Harvard University (Other); Baylor College of Medicine (Other); Dana-Farber Cancer Institute (Other); University of Washington (Other); Fred Hutchinson Cancer Center (Other); Johns Hopkins University (Other); Mayo Clinic (Other); M.D. Anderson Cancer Center (Other); Northwestern University (Other); University of Michigan (Other); University of California, San Francisco (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 07-053
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue, serum, plasma, and lymphocytes

GROUPS / COHORTS (2):
- 1: patients scheduled to receive standard of care with a Radical prostatectomy
  Interventions: Other: Questioners, blood specimens, prostate tissue specimens
- 2: patients scheduled to receive standard of care with radiation therapy
  Interventions: Other: Questioners, blood specimens, prostate tissue specimens

INTERVENTIONS:
Other: Questioners, blood specimens, prostate tissue specimens — You will be asked to fill out a confidential questionnaire asking for information such as medical history, family history of cancer, and potential exposures.
  Each patient will provide 7 unstained paraffin sections from prostate biopsies, one tube of blood for serum, and one tube for plasma and buffy coat.
  Groups: 1
Other: Questioners, blood specimens, prostate tissue specimens — You will be asked to fill out a confidential questionnaire asking for information such as medical history, family history of cancer, and potential exposures.
  Each patient will provide 7 unstained paraffin sections from prostate biopsies, one tube of blood for serum, and one tube for plasma and buffy coat.
  Groups: 2

SUMMARY:
Radical Prostatectomy (removal of the prostate) or radiation therapy provide excellent outcomes for patients with localized (confined to one area) disease, yet there is still no effective treatment once the disease has spread beyond the prostate gland. Typically, a serum PSA test is done to diagnose prostate cancer. Following diagnosis, a prostate biopsy and other tests help to classify the patient's disease according to the likelihood of a recurrence. However, these assessments are imperfect. There is a need to identify and evaluate prostate biomarkers that will provide exact information regarding the likelihood of a recurrence (prediction) of prostate cancer.

DETAILED DESCRIPTION:
The Inter-SPORE Prostate Biomarkers Study (IPBS) was established to prospectively collect and analyze biological specimens to predict and validate outcomes after treatment for prostate cancer. The study population will consist of patients scheduled to receive standard of care therapy for localized prostate cancer, either radical prostatectomy (RP) or radiation therapy (XRT; includes external beam radiation, brachytherapy, or both). Seven hundred (700) patients (350 RP, 350 XRT) will be recruited from 11 SPORE sites over a two-year interval. We will collect serum, plasma, lymphocytes, and prostate tissue samples for distribution to collaborating biomarker validation sites at other prostate SPOREs, along with clinical and epidemiologic data.

ELIGIBILITY:
Inclusion Criteria:

* Males, 35 years of age or older, with histologically confirmed prostate adenocarcinoma, that is clinically localized to the prostate gland.
* Biopsy performed at the SPORE institution.
* No prior therapy for prostate cancer (patients who receive neoadjuvant therapy after collection of blood and biopsy samples are eligible).
* The patient should have 2 or more cores involved with carcinoma. The minimum amount of tumor submitted should be 5 mm, or at least 40% of the core involved with tumor. (This amount can be made up from 2 positive cores if 1 core is insufficient).
* Patients with clinical stage T1-T2a NXM0 prostate cancer who elect to be treated with RP or XRT (includes external beam radiation, brachytherapy, or both) at the SPORE institution.
* Patients with a nomogram predicted 5-year probability of freedom from biochemical recurrence (Kattan 1998) of less than or equal to 85% (patients with intermediate risk of recurrence).
* Ability and willingness to sign informed consent

Exclusion Criteria:

* Participation in a therapeutic clinical trial with an experimental agent.
* Previous cancer of any kind except non-melanoma skin cancer
* Previous surgical or minimally invasive treatment for enlarged prostate (e.g. TURP, TUNA, TUIP, laser, microwave)
* Use of anti-androgen drugs during the 6 months prior to diagnosis
* Use of 5-alpha-reductase inhibitors during the 6 months prior to diagnosis

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 11 cancer centers in the USA
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Coll & contrib bio spec to Inter-SPORE Prostate Biomarker Study men with clinical localized prostate ca sched to get standard of care therapy for localized prost ca, either radical prostatectomy, RT therapy | pre-treatment and at yearly intervals during follow-up.

SECONDARY OUTCOMES:
To participate in the IPBS by conducting a prospective analysis of the prognostic utility of serum hK2 in predicting biochemical recurrence after definitive local therapy for prostate cancer. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org